CLINICAL TRIAL: NCT03642353
Title: Triclosan as Adjunctive Therapy in the Plaque Control in Children From Generalized Aggressive Periodontitis Families. A Controlled and Randomized Clinical Trial.
Brief Title: Triclosan as Adjunctive Therapy in the Plaque Control in Children From Generalized Aggressive Periodontitis Families.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Principal Investigator, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 103/2015
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Generalized Aggressive Periodontitis
Keywords: plaque control; bacteria; inflammation; familial aggregation; prevention
MeSH Terms: conditions — Inflammation | interventions — Triclosan; Toothpastes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- G1: Triclosan/health children (Experimental): Children from health parents will use the triclosan toothpaste for 45 days.
  Interventions: Drug: Triclosan
- G2: Placebo/health children (Placebo Comparator): Children from health parents will use the placebo toothpaste for 45 days.
  Interventions: Drug: Placebo
- G3: Triclosan/GAP children (Experimental): Children from GAP parents will use the triclosan toothpaste for 45 days.
  Interventions: Drug: Triclosan
- G4: Placebo/GAP children (Placebo Comparator): Children from GAP parents will use the placebo toothpaste for 45 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Triclosan — Children will be included in a cross-over study with control of plaque using Triclosan/placebo toothpaste for 4 months. Each child will be tested for placebo toothpaste for 45 days and for Triclosan toothpaste for more 45 days. At the beginning of each test, they will be included in a washout period with placebo toothpaste for 15 days.
  Other Names: Colgate Total Advanced Toothpaste
  Arms: G1: Triclosan/health children; G3: Triclosan/GAP children
Drug: Placebo — Children will be included in a cross-over study with control of plaque using Triclosan/placebo toothpaste for 4 months. Each child will be tested for placebo toothpaste for 45 days and for Triclosan toothpaste for more 45 days. At the beginning of each test, they will be included in a washout period with placebo toothpaste for 15 days.
  Other Names: Colgate Cavity Protection 0.76 % Toothpaste
  Arms: G2: Placebo/health children; G4: Placebo/GAP children

SUMMARY:
Generalized aggressive periodontitis (GAP) is an inflammatory disease that causes the severe and rapid destruction of periodontal tissue. A relatively constant microbiological pattern, an altered inflammatory condition and familial aggregation of cases were described as important characteristics of this disease. In this vein, studies evaluating children of GAP patients were made and identified early microbiological and inflammatory alterations in this population, suggesting that these factors could favor the disease development. Thus, the aim of this project is to evaluate if the use of toothpaste with Triclosan could have a beneficial effect in control the microbiota and the inflammatory condition in children from parents with GAP, comparing them to children of periodontally healthy parents. 20 children (6-12 years old) from GAP parents and 20 children (6-12 years old) from periodontally healthy parents will be selected and will participate in a cross-over placebo study. All children will be included in a 15-day period of control of plaque to standardize the hygiene technique using only the placebo toothpaste. After this period, the children will be divided randomly into 4 groups: G1: Triclosan/health children; G2: Placebo/health children; G3: Triclosan/GAP children; G4: Placebo/GAP children and they will use the specific paste described for each group for 45 days. After this period, all children will repeat the 15 days interval, using only the placebo toothpaste, to remove the Triclosan effect and to standardize the oral hygiene again. Posteriorly, the crossing of groups will be done and children will be reallocated to change the used toothpaste. Thus, children that were in G1 will be reallocated in G2, children of G2 will be reallocated in G1, children of G3 will be in G4 and children of G4 will be in G3, staying in this new group for more 45 days. The evaluated periods will be baseline, 15 days, 30 days and 45 days while children stay in G1, G2, G3 or G4. In these periods children will be clinically evaluated for the periodontal parameter and sample collection of crevicular gingival fluid (GCF) and subgingival biofilm from incisors and molars will be done. Luminex/MAGpix technology will be used to detect IL-1β, IL-4, IL-6, IL-8, IL-10, IL-17, TNF-α, INF-γ in the GCF. The subgingival biofilm will be used to evaluate the Porphyromonas gingivalis, Tannerella forsythia, Aggregatibacter actinomycetemcomitans levels by real-time PCR.

DETAILED DESCRIPTION:
The data from each group will be compared by Student's t-test, Mann-Whitney test and chi-square test and a correlation between the inflammatory markers level and the subgingival bacterial concentration will be evaluated by Spearman's correlation and regression analysis. The significance level for all analysis will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Present parents diagnosed with periodontal health or generalized aggressive periodontitis
* Present between 6 and 12 years old
* Present good general health

Exclusion Criteria:

* The use of antibiotics or anti-inflammatories 6 months before the beginning of the study.
* Any Any change in the child's motor condition that interferes with the performance of appropriate hygiene procedures.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01-30 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Change of the baseline bledding on probing at 45 days | Baseline and 45 days for each test
  Bleeding induced at the depth of the gingival sulcus or periodontal pocket after probing

SECONDARY OUTCOMES:
Change of the baseline plaque index at 45 days | Baseline and 45 days for each test
  Reduction in the amount of plaque accumulation around the gingival marginal after the therapy.
Change of the baseline inflamatory markers levels in gingival crevicular fluid (pg/uL) at 45 days | Baseline and 45 days for each test
  Concentration of IL-1β, IL-4, IL-6, IL-8, IL-10, IL-17, TNF-α and INF-γ released in gingival crevicular fluid
Change in the Microbial composition at 45 days | Baseline and 45 days for each test
  Concentration of bacteria in the subgingival biofilm

CONTACTS AND LOCATIONS:
Overall Officials: Renato CV Casarin, Prof. Dr., Study Chair — University of Campinas, UNICAMP
Locations (1):
- University of Campinas, UNICAMP, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Monteiro MF, Tonelli H, Reis AA, Casati MZ, Silverio KG, Nociti Junior FH, Sallum EA, Casarin RCV. Triclosan toothpaste as an adjunct therapy to plaque control in children from periodontitis families: a crossover clinical trial. Clin Oral Investig. 2020 Apr;24(4):1421-1430. doi: 10.1007/s00784-019-03121-6. Epub 2020 Jan 6. PMID 31907625